CLINICAL TRIAL: NCT00546559
Title: Differential Metabolic Effects of Statins
Status: Completed | Type: Observational
Sponsor: Gachon University Gil Medical Center (Other)
Other Study IDs: GMC-200406
Record Dates: First submitted 2007-10-18; First posted 2007-10-19 (Estimated); Last update posted 2008-08-29 (Estimated); Status verified 2008-08

CONDITIONS: Hypercholesterolemia
Keywords: Lipophilic statins; Insulin resistance; simvastatin and pravastatin may have differential metabolic effects in hypercholesterolemic patients.
MeSH Terms: conditions — Hypercholesterolemia; Insulin Resistance | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Simvastatin; Pravastatin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: statins (simvastatin, pravastatin)

SUMMARY:
The investigators hypothesized simvastatin and pravastatin may have differential metabolic effects in hypercholesterolemic patients.

ELIGIBILITY:
Inclusion Criteria:

* Low-density lipoprotein cholesterol levels > 130

Exclusion Criteria:

* Overt liver disease,
* Chronic renal failure
* Hypothyroidism
* Myopathy
* Uncontrolled diabetes
* Severe hypertension

Ages: 25 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2004-01; Study Completion 2008-03

PRIMARY OUTCOMES:
Simvastatin and pravastatin may have differential metabolic effects in hypercholesterolemic patients.

CONTACTS AND LOCATIONS:
Overall Officials: Kwang K Koh, MD,PhD, Principal Investigator — Gachon University Gil Medical Center
Locations (1):
- Gil Medical Center, Incheon, South Korea

REFERENCES:
- [Result] Yada T, Nakata M, Shiraishi T, Kakei M. Inhibition by simvastatin, but not pravastatin, of glucose-induced cytosolic Ca2+ signalling and insulin secretion due to blockade of L-type Ca2+ channels in rat islet beta-cells. Br J Pharmacol. 1999 Mar;126(5):1205-13. doi: 10.1038/sj.bjp.0702397. PMID 10205010